CLINICAL TRIAL: NCT07048587
Title: Evaluating the Diagnostic Efficacy of β-hCG Levels in Uterine Cavity Lavage: A Potential Tool for Identifying Pregnancies of Unknown Location (PUL) and Ectopic Pregnancies
Brief Title: Beta-HCG Levels in Uterine Cavity Lavage for Pregnancies of Unknown Location
Acronym: BHCG-UCL-DEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Reyyan Gokcen Iscan, Consultant gynecologist and obstetrician, MD, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-101
Record Dates: First submitted 2025-05-07; First posted 2025-07-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy, Ectopic; Early Pregnancy Loss
Keywords: ectopic pregnancy, beta-hCG, early pregnancy loss, uterine cavity lavage
MeSH Terms: conditions — Pregnancy, Ectopic; Abortion, Spontaneous | interventions — Diagnosis, Differential

STUDY DESIGN:
Intervention Model Description: This prospective study aims to evaluate the diagnostic potential of beta-hCG levels in uterine cavity lavage fluid for differentiating between ectopic pregnancy and early pregnancy loss. The study includes female patients aged 18-45 with positive serum beta-hCG, inconclusive diagnoses, and abnormal beta-hCG progression. Participants undergo uterine cavity lavage before scheduled probe curettage, with 5 cc of saline solution administered and 3 cc of aspirated liquid collected for beta-hCG measurement. Before the intervention beta-hCG is measured in venous blood.Data collection involves beta-hCG levels from lavage fluid, pathology results from curettage, and final diagnoses. Analysis compares lavage fluid beta-hCG levels with pathology results and final diagnoses to determine a potential cut-off value for differentiation. Outcome measures include diagnostic accuracy, correlation between lavage fluid beta-hCG levels and final diagnoses, and sensitivity/specificity of the proposed method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm; Patients with a β-hCG level of 1500-2000 mIU/mL with pregnancy of unknown location (Experimental): The study arm includes patients aged 18-45 with positive serum β-hCG and unclear clinical or ultrasound results. On the day of the intervention, a blood sample is collected to measure β-hCG levels, followed by the irrigation of the uterine cavity with 5 ml prior to the probe curettage (P/C).Three ml of wash fluid is collected for β-hCG measurement. After collecting the uterine lavage fluid samples, each specimen was frozen at -80 ºC and then all samples analyzed later, on the same day.
  Interventions: Diagnostic Test: Beta-hCG levels in the uterine cavity lavage for differential diagnosis in pregnancy of unknown locations and ectopic pregnancy

INTERVENTIONS:
Diagnostic Test: Beta-hCG levels in the uterine cavity lavage for differential diagnosis in pregnancy of unknown locations and ectopic pregnancy — The intervention in this study centers on utilizing beta-hCG levels in uterine cavity lavage as a diagnostic tool to differentiate between ectopic pregnancy and early pregnancy loss.The procedure includes females aged 18-45 with positive serum beta-hCG, inconclusive clinical findings, and transvaginal ultrasound results, focusing on beta-hCG levels below 1500-2000 mIU/mL and abnormal progression.The intervention performed before probe curettage (P/C). Before the intervention beta-hCG is measured in venous blood. Patients undergo uterine cavity lavage with 5 ml of saline solution administered and 3 ml of aspirated liquid collected for beta-hCG measurement. Data collection involves beta-hCG levels from lavage fluid and venous blood, pathology results.After the samples were collected, each one was frozen at -80 ºC. All uterine lavage samples were then analyzed later on the same day.

SUMMARY:
The goal of this interventional study is to investigate the role of beta-hCG levels in uterine cavity lavage for differentiating between ectopic pregnancy and early pregnancy loss in female patients aged 18-45 years. The main questions it aims to answer are as follows:

1. Can beta-hCG levels in uterine cavity lavage provide a decisive cut-off value for distinguishing between ectopic pregnancy and intrauterine pregnancy (early pregnancy loss)?
2. How do beta-hCG levels in uterine cavity lavage compare with venous blood beta-hCG levels and pathological results, final diagnoses?

Researchers will compare beta-hCG levels in uterine cavity lavage to pathological results and final diagnoses to determine whether this method can provide a quick and accurate differentiation between ectopic pregnancy and early pregnancy loss.

Participants will:

* Undergo uterine cavity lavage with 5 cc of saline solution before anesthesia and probe curettage
* Have 3 cc of aspirated liquid collected in a gel tube for beta-hCG level measurement
* Proceed with the scheduled probe curettage procedure

The study focuses on patients with positive serum beta-hCG values, serum beta-hCG levels below the differential level (<1500-2000 mIU/mL), abnormal beta-hCG progression in consecutive measurements, and inconclusive transvaginal ultrasound results for differential diagnosis.

DETAILED DESCRIPTION:
This study aims to investigate the potential of using beta-hCG levels in uterine cavity lavage as a diagnostic tool for differentiating between ectopic pregnancy and early pregnancy loss. The research focuses on female patients aged 18-45 years who present with positive serum beta-hCG values but inconclusive clinical findings and transvaginal ultrasound results.

The study will specifically target patients with serum beta-hCG levels below the differential level (typically <1500-2000 mIU/mL) and abnormal beta-hCG progression in consecutive measurements. These patients, who are scheduled for probe curettage (P/C), will undergo uterine cavity lavage prior to the procedure.

The lavage process involves administering 5 cc of saline solution into the uterine cavity before anesthesia and the P/C procedure. Subsequently, 3 cc of the aspirated liquid will be collected in a gel tube for beta-hCG level measurement.

The primary objective is to determine if there is a decisive cut-off value in the beta-hCG levels of the lavage fluid that can accurately differentiate between ectopic pregnancy and early pregnancy loss. This approach aims to provide a quick and minimally invasive diagnostic method, potentially reducing the need for more invasive procedures or operations.

The results of the beta-hCG measurements from the lavage fluid will be compared with the pathology results from the P/C and the final diagnosis. This comparison will help evaluate the accuracy and reliability of this novel diagnostic approach.

If successful, this method could offer a faster and less invasive way to distinguish between ectopic pregnancy and early pregnancy loss in cases where current diagnostic methods are inconclusive. This could potentially lead to earlier and more appropriate interventions, improving patient care and outcomes in early pregnancy complications.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45
* Beta-HCG positivity
* Hemodynamically stable
* Consecutive beta-hCG measurements do not show a normal pregnancy,
* Beta-hCG is below the differential level (<1500-2000 mIU / mL) and TV-USG examination is insufficient for differential diagnosis

Exclusion Criteria:

* Hemodynamic instability
* Confirmed intrauterine pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with Reproductive Age
Enrollment: 121 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Comparison of beta-hCG levels in simultaneously collected uterine lavage and venous blood with pathology results | The time frame from patient enrollment in the intervention to the receipt of pathology results and comparison with intrauterine lavage results was an average of three weeks.
  Primary outcome include diagnostic accuracy, correlation between lavage fluid and venous blood beta-hCG levels and final diagnoses.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Women and Children Diseases Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Will be shared after complitation of primary outcomes